CLINICAL TRIAL: NCT06851286
Title: The Effect of Laughter Therapy Given to Mothers in The Postpartum Period on Their Perceived Stress, Sleep Quality and Breastfeeding Self-Efficacy Level; Randomized Controlled Trial
Brief Title: Effects of Laughter Therapy on Postpartum Mothers' Stress, Sleep, and Breastfeeding
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Havva Tokgöz Kekeç, PhD Student, Msc Midwife, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024/616; Researcher (Other: Selçuk University)
Record Dates: First submitted 2025-02-16; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Postnatal Care; Lactation
Keywords: Sleep Quality; Breastfeeding Self-Efficacy Level; Laughter Therapy; Perceived Stress
MeSH Terms: conditions — Breast Feeding; Sleep Initiation and Maintenance Disorders | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: After randomization is achieved, a WhatsApp group will be established with the mothers in the laughter therapy group. Before starting the application, the "Zoom" program will be downloaded to the phones or computers of the mothers in the laughter therapy group. Afterwards, an online application will be carried out in groups via Zoom, by determining a common day and time according to the working hours of the mothers and the researcher. Groups will be formed with at least 5-10 people, and laughter therapy will be applied to the groups for 4 weeks, 2 sessions per week, for a total of 8 sessions. No intervention will be made to the control group, and they will be asked to fill out the survey forms simultaneously. A laughter yoga session; It is approximately 30 minutes and consists of four parts. These sections; hand clapping and warm-up exercises, deep breathing exercises, childish games and laughter exercises.
Who Masked: Participant, Outcomes Assessor
Masking Description: In the study, the process of assigning mothers to the laughter therapy and control groups was done by simple randomisation to ensure similarity between the groups. To ensure randomisation in the study, a table of random numbers was created by dividing into two groups according to the number determined on https://www.randomizer.org/. Two random number series (set 1 and set 2) between 1- 120 were created in the system using the Random Integer Generator method in the Numbers subheading of this site. The 120 women who met the inclusion criteria were assigned to 60 laughter therapy groups and 60 control groups in a 1:1 ratio by simple randomisation method. Which group was the intervention or control group was determined by drawing lots at the beginning of the study. The mothers included in the study did not know which group they were in at first. After the individuals who met the inclusion criteria and volunteered to participate in the study were determined, the participants were assigned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laughter therapy group (Experimental): After randomization is achieved, a WhatsApp group will be established with the mothers in the laughter therapy group. Before starting the application, the "Zoom" program will be downloaded to the phones or computers of the mothers in the laughter therapy group. Afterwards, an online application will be carried out in groups via Zoom, by determining a common day and time according to the working hours of the mothers and the researcher. Groups will be formed with at least 5-10 people, and laughter therapy will be applied to the groups for 4 weeks, 2 sessions per week, for a total of 8 sessions.
  Interventions: Behavioral: Laughter Therapy
- control group (No Intervention): No intervention will be made to the control group, they will be asked to fill out the survey forms simultaneously.

INTERVENTIONS:
Behavioral: Laughter Therapy — A laughter yoga session; It is approximately 30 minutes and consists of four parts. These sections; hand clapping and warm-up exercises, deep breathing exercises, childish games and laughter exercises. In each laughter yoga session, the first three parts are the same, but the laughter exercises in the fourth part vary. In the first session of each new group, the introduction of laughter yoga, its purpose and objectives will be discussed. 10 minutes will be allocated for this section in the first session of each group. Therefore, the first session is planned to be 40 minutes in each group and all subsequent sessions are planned to be 30 minutes.
  Arms: laughter therapy group

SUMMARY:
Postnatal period is an important developmental transition period for women. Stress in the postnatal period is one of the most common mental health problems and most mothers report experiencing stress in the perinatal period. In addition, stress and negative mental health also threaten breastfeeding self-efficacy. The postnatal period is an important stage in terms of early initiation and maintenance of breastfeeding. Breastfeeding self-efficacy is a mother's perceived confidence in her ability to breastfeed her newborn baby. Therefore, midwives are expected to assess women and identify women in need of supportive interventions and consciously contribute to their treatment. Another common problem in the postnatal period is poor sleep quality. It was determined that an increase in sleep quality and perceived social support positively affected breastfeeding self-efficacy of postpartum women. In addition, poor sleep quality poses a threat for negative mental health outcomes for women in the postpartum period. Previous studies reflect mothers' desire for non-pharmacological interventions and a high degree of satisfaction with these therapies. Laughter therapy, one of the main non-pharmacological interventions, is recognised as a universal approach to reduce stress and anxiety. The postnatal period is a fragile period with physical and psychological changes as well as hormonal changes in the mother. Poor mental health of the mother poses a danger to the well-being of the mother and the baby. Mothers in the postpartum period need low-cost, easily accessible preventive interventions to prevent these problems. In this context, the aim of this study is to determine the effect of laughter therapy given to mothers in the postpartum period on perceived stress, sleep quality and breastfeeding self-efficacy level in mothers.

DETAILED DESCRIPTION:
The postnatal period is an important developmental transition period for women and mothers experience various difficulties. Therefore, midwives are expected to assess women and identify women in need of supportive interventions and consciously contribute to their treatment. Previous studies reflect mothers' desire for non-pharmacological therapies and a high degree of satisfaction with these therapies. Laughter therapy, one of the main non-pharmacological interventions, is recognised as a universal approach to reduce stress and anxiety. Laughter therapy is a new, simple, cost-effective, non-invasive, non-invasive, widely available online, easily accessible and effective method. Laughter therapy has been applied to many different patient populations and healthy individuals in a variety of settings, and studies have reported benefits such as improved sleep quality, decreased depression, pain and stress hormones, improved mood and life satisfaction, increased prenatal attachment and breastfeeding self-efficacy. These benefits document the positive role of laughter therapy in improving the quality of life of individuals. Laughter therapy is a type of cognitive-behavioural therapy that can improve physical, psychological and ultimately quality of life. Laughter therapy can be used for both preventive and therapeutic purposes. In contrast, the negative effects of laughter and humour are negligible.

In conclusion, laughter is a human and universal value. Using laughter effectively to improve well-being and facilitate adaptation to the changes experienced in this period can significantly improve quality of life. Mothers in the postpartum period need low-cost, easily accessible preventive interventions to prevent these problems. However, to achieve this, health professionals need to be aware of the most appropriate evidence-based interventions. The number of studies investigating the effect of laughter therapy on women's health is limited in Turkey. In order to increase evidence-based data, there is a need to investigate the potential effectiveness of laughter therapy interventions in terms of women's health. In this context, the aim of this study was to determine the effect of laughter therapy given to mothers in the postnatal period on perceived stress, sleep quality and breastfeeding self-efficacy level. It is thought that the results of this study will guide midwives to be aware of the effectiveness of laughter therapy and to plan interventions to improve the quality of life of mothers.

ELIGIBILITY:
Inclusion Criteria:

* At least primary school graduate
* Over the age of 18
* Those who volunteer to participate in the research
* Heterosexual
* Having a single and healthy baby
* Postpartum 1-12 month old baby
* Women who can use Zoom program

Exclusion Criteria:

* Those who do not speak Turkish,
* Those with hearing and visual impairments,
* Those with mental disabilities,
* Those diagnosed with a known psychiatric disease,
* Mothers who do not breastfeed
* Mothers who have babies with disabilities and chronic health problems
* Women with physical conditions that prevent them from participating in laughter yoga sessions (respiratory distress, persistent cough, vertiligo, severe heart disease, hemorrhoids, any type of hernia such as neck, waist or inguinal hernia, severe back pain, urinary incontinence, epilepsy, etc.),
* Women who use medication or use another non-pharmacological method to reduce stress.

Women who develop an acute health problem in themselves or their babies, who have a sudden hospitalisation of the mother or baby, mothers who lose their babies, women who do not attend all of the laughter therapy sessions and women who cannot be reached after the application will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — breastfeeding mothers in the postpartum period
Enrollment: 120 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale | 1st Time: Day 1, 2nd Time: Day 30, 3rd Time: Day 60
  It was developed by Cohen, Kamarck & Mermelste (1983), and in the reliability study, the Cronbach Alpha value was found to be 0.86. The Cronbach Alpha value of the "Perceived Stress Scale", which was adapted into Turkish by Bilge, Öğce, Genç and Oran (2007) and whose validity and reliability studies were conducted, was found to be 0.81. Three items of the scale, prepared in a 5-point Likert type (0 never, 4 very often), are reverse-worded (items 4, 5, 6), and five items are literal (items 1, 2, 3, 7, and 8). A total score of 0-32 is taken from the scale. It has two subscales: perceived stress (items 1, 2, 3, 7, 8) and perceived coping (items 4, 5, and 6). The scale is evaluated on both total score and subscale scores. A high total score means a high perceived stress level. High scores from the subscales are a negative situation.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 1st Time: Day 1, 2nd Time: Day 30, 3rd Time: Day 60
  The PSQI was developed by Buysse et al. (1989) (20) and its Turkish validity and reliability was performed by Ağargün et al. (1996). The PSQI provides information about sleep quality in the last month and the type and severity of sleep disturbance. In the scale consisting of 24 questions in total, 18 questions are scored. The scale consists of 7 sub-dimensions that provide information about the individual's 'Subjective Sleep Quality', 'Sleep Latency', 'Sleep Duration', 'Habitual Sleep Efficiency', 'Sleep Disorder', 'Sleep Medication Use' and 'Daytime Dysfunction'. Each sub-dimension is evaluated on a 0-3 point scale (item 0=no distress, 3=serious distress). The total score of all sub-dimensions gives the total score of the scale (min- max=0-21). Sleep quality is classified as good between 0-4 points and poor sleep quality between 5-21 points.

OTHER OUTCOMES:
Breastfeeding Self-Efficacy Scale | 1st Time: Day 1, 2nd Time: Day 30, 3rd Time: Day 60
  In 2003, a 14-item short form of the 33-item scale developed by Dennis and Faux was developed to assess mothers' breastfeeding self-efficacy levels. Tokat Aluş and Okumuş (2010) conducted a Turkish reliability and validity study of the short form of the Breastfeeding Self-Efficacy Scale and found that it was suitable for Turkish culture. The Breastfeeding Self-Efficacy Short Form Scale is a 5-point Likert-type scale (1=Never sure and 5=Always sure). The minimum score that can be obtained from the scale is 14 and the maximum score is 70. The higher the score, the higher the breastfeeding self-efficacy. The average administration time of the scale is 5-7 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Selçuk University Faculty of Medicine Hospital, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Akın, B., Tanyer, D. (2021). SPIRIT 2013 Bildirisi: Klinik Deneyler İçin Standart Protokol Maddelerinin Tanımlanması. HUHEMFAD, 8(1):117-2.
- [Result] Boutron I, Altman DG, Moher D, Schulz KF, Ravaud P; CONSORT NPT Group. CONSORT Statement for Randomized Trials of Nonpharmacologic Treatments: A 2017 Update and a CONSORT Extension for Nonpharmacologic Trial Abstracts. Ann Intern Med. 2017 Jul 4;167(1):40-47. doi: 10.7326/M17-0046. Epub 2017 Jun 20. PMID 28630973
- [Result] Zhao J, Yin H, Zhang G, Li G, Shang B, Wang C, Chen L. A meta-analysis of randomized controlled trials of laughter and humour interventions on depression, anxiety and sleep quality in adults. J Adv Nurs. 2019 Nov;75(11):2435-2448. doi: 10.1111/jan.14000. Epub 2019 May 9. PMID 30882915
- [Result] Yim J. Therapeutic Benefits of Laughter in Mental Health: A Theoretical Review. Tohoku J Exp Med. 2016 Jul;239(3):243-9. doi: 10.1620/tjem.239.243. PMID 27439375
- [Result] Werner-Bierwisch T, Pinkert C, Niessen K, Metzing S, Hellmers C. Mothers' and fathers' sense of security in the context of pregnancy, childbirth and the postnatal period: an integrative literature review. BMC Pregnancy Childbirth. 2018 Dec 4;18(1):473. doi: 10.1186/s12884-018-2096-3. PMID 30509217
- [Result] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575
- [Result] van der Wal CN, Kok RN. Laughter-inducing therapies: Systematic review and meta-analysis. Soc Sci Med. 2019 Jul;232:473-488. doi: 10.1016/j.socscimed.2019.02.018. Epub 2019 Mar 5. PMID 31029483
- [Result] Stremler, R., Sharkey, K.M., & Wolfson, A.R. (2017). Postpartum period and early motherhood. In M. Kryger, T. Roth, &W. Dement (Eds.), Principles and practice of sleep medicine (6th ed., pp. 1547Y1552). Philadelphia, PA: Elsevier.
- [Result] Pierce M, Hope HF, Kolade A, Gellatly J, Osam CS, Perchard R, Kosidou K, Dalman C, Morgan V, Di Prinzio P, Abel KM. Effects of parental mental illness on children's physical health: systematic review and meta-analysis. Br J Psychiatry. 2020 Jul;217(1):354-363. doi: 10.1192/bjp.2019.216. PMID 31610824
- [Result] Okun ML, Mancuso RA, Hobel CJ, Schetter CD, Coussons-Read M. Poor sleep quality increases symptoms of depression and anxiety in postpartum women. J Behav Med. 2018 Oct;41(5):703-710. doi: 10.1007/s10865-018-9950-7. Epub 2018 Jul 20. PMID 30030650
- [Result] Namazinia M, Mazlum SR, Mohajer S, Lopez V. Effects of laughter yoga on health-related quality of life in cancer patients undergoing chemotherapy: a randomized clinical trial. BMC Complement Med Ther. 2023 Jun 12;23(1):192. doi: 10.1186/s12906-023-04028-2. PMID 37303065
- [Result] Moon H, Journ S, Lee S. Effect of Laughter Therapy on Mood Disturbances, Pain, and Burnout in Terminally Ill Cancer Patients and Family Caregivers. Cancer Nurs. 2024 Jan-Feb 01;47(1):3-11. doi: 10.1097/NCC.0000000000001162. Epub 2022 Dec 11. PMID 36066344
- [Result] Meier M, Wirz L, Dickinson P, Pruessner JC. Laughter yoga reduces the cortisol response to acute stress in healthy individuals. Stress. 2021 Jan;24(1):44-52. doi: 10.1080/10253890.2020.1766018. Epub 2020 May 26. PMID 32393092
- [Result] Küçükkelepçe, D. Ş., Ünver, H., & Kurt, N. (2024). Kahkaha Yogasının Emzirme Öz-Yeterliliği Üzerine Etkisinin İncelenmesi: Randomize Kontrollü Çalışma. Journal of Academic Research in Nursing, 10(1), 57-66. https://doi.org/10.55646/jaren.2024.93064
- [Result] Konukbay D, Oksuz E, Guvenc G. Breastfeeding self-efficacy in terms of sleep quality, perceived social support, depression and certain variables: a cross-sectional study of postpartum women in Turkey. BMC Pregnancy Childbirth. 2024 Apr 2;24(1):231. doi: 10.1186/s12884-024-06456-5. PMID 38566031
- [Result] Ko Y, Park S. A pilot randomized controlled trial of distance laughter therapy for mothers' level of depression, anxiety, and parental stress during the COVID-19 pandemic. PLoS One. 2023 Jul 14;18(7):e0288246. doi: 10.1371/journal.pone.0288246. eCollection 2023. PMID 37450484
- [Result] Khadka R, Hong SA, Chang YS. Prevalence and determinants of poor sleep quality and depression among postpartum women: a community-based study in Ramechhap district, Nepal. Int Health. 2020 Feb 12;12(2):125-131. doi: 10.1093/inthealth/ihz032. PMID 31294785
- [Result] Henrique AJ, Gabrielloni MC, Rodney P, Barbieri M. Non-pharmacological interventions during childbirth for pain relief, anxiety, and neuroendocrine stress parameters: A randomized controlled trial. Int J Nurs Pract. 2018 Jun;24(3):e12642. doi: 10.1111/ijn.12642. Epub 2018 Mar 7. PMID 29512230
- [Result] Harputlu D, Ozturk FO, Aydin D, Akyol C, Tezel A. Effect of Laughter Yoga on Sleep and Quality of Life in Individuals With Fecal Ostomies: A Randomized Controlled Trial. J Wound Ostomy Continence Nurs. 2023 Jul-Aug 01;50(4):307-312. doi: 10.1097/WON.0000000000000988. PMID 37467409
- [Result] Dominguez-Solis E, Lima-Serrano M, Lima-Rodriguez JS. Non-pharmacological interventions to reduce anxiety in pregnancy, labour and postpartum: A systematic review. Midwifery. 2021 Nov;102:103126. doi: 10.1016/j.midw.2021.103126. Epub 2021 Aug 14. PMID 34464836
- [Result] Dennis CL, Faux S. Development and psychometric testing of the Breastfeeding Self-Efficacy Scale. Res Nurs Health. 1999 Oct;22(5):399-409. doi: 10.1002/(sici)1098-240x(199910)22:53.0.co;2-4. PMID 10520192
- [Result] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Result] Christian LM, Carroll JE, Porter K, Hall MH. Sleep quality across pregnancy and postpartum: effects of parity and race. Sleep Health. 2019 Aug;5(4):327-334. doi: 10.1016/j.sleh.2019.03.005. Epub 2019 May 20. PMID 31122875
- [Result] Cattarius BG, Schlarb AA. How the Sleep of Couples Changes from Pregnancy to Three Months Postpartum. Nat Sci Sleep. 2021 Feb 24;13:251-261. doi: 10.2147/NSS.S259072. eCollection 2021. PMID 33658879
- [Result] Bilge A., F, Öğce., Genç, R. E., Oran, N.T. (2009). Algılanan Stres Ölçeği (ASÖ)'nin Türkçe Versiyonunun Psikometrik Uygunluğu, Ege Üniversitesi Hemşirelik Yüksekokulu Dergisi, 2(25), 61-72, 2009.
- [Result] Alus Tokat M, Okumus H, Dennis CL. Translation and psychometric assessment of the Breast-feeding Self-Efficacy Scale-Short Form among pregnant and postnatal women in Turkey. Midwifery. 2010 Feb;26(1):101-8. doi: 10.1016/j.midw.2008.04.002. Epub 2008 Jun 9. PMID 18541350
- [Result] Agapinar Sahin S, Bekar M. The influence of laughter yoga on pregnancy symptoms, mental well-being, and prenatal attachment: A randomized controlled study. Health Care Women Int. 2023 Jun;44(6):782-801. doi: 10.1080/07399332.2022.2164284. Epub 2023 Jan 10. PMID 36625775